CLINICAL TRIAL: NCT02978963
Title: Cognitive Behavioral Therapy for Adolescents With Excessive Worry - a Case Series
Brief Title: CBT for Adolescents With Excessive Worry
Acronym: BiPOro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Serlachius, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN DNR 2016/1408-31/5
Record Dates: First submitted 2016-11-13; First posted 2016-12-01 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Excessive Worry
Keywords: Excessive worry; Worry; Adolescents; Intolerance of uncertainty
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): All participants will receive cognitive behavioral therapy for excessive worry. Focus in treatment will be on reducing participants' intolerance uncertainty through in vivo and imaginary exposure to uncertainty inducing situations and thoughts. Treatment will also contain psycho education about anxiety and worry, as well as planning for maintenance of treatment gains. Parents of the participants will receive support and education about worry through an internet-delivered program.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — CBT focused on reducing intolerance of uncertainty
  Other Names: CBT

SUMMARY:
This case series aims to test the feasibility and acceptability of streamlined cognitive behavioral therapy (CBT) for adolescents with excessive worry. The treatment protocol focuses on reducing intolerance of uncertainty and the hypothesis is that this will help reduce worry.

DETAILED DESCRIPTION:
This pilot study aims to test a new form of Cognitive Behavioral Therapy for adolescents with excessive worry. The investigators will include 12 participants with excessive worry and test the treatment which focuses on reducing intolerance of uncertainty (IU) in order to reduce worry.

Participants will be randomized to either one, two or three weeks of weekly baseline measurements prior to starting treatment, and will thus work as their on controls in this case series design.

Primary outcome measures will be collected at 12 weeks after treatment start. Participants will be followed up at three months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* A score on PSWQ-C of at least 22
* Age between 13 and 17 years
* Ability to read and write in Swedish
* A parent or caregiver that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* Diagnosis of autism spectrum disorder, psychosis, bipolar disorder or severe eating disorder
* Present risk of suicide
* Ongoing substance dependence
* Occurrence of domestic violence
* Completed CBT for any anxiety disorder within the last 6 months (defined as at least 5 sessions of CBT including in vivo exposure sessions)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire for Children (PSWQ-C) | At 12 weeks after treatment starts
  Child and parent version

SECONDARY OUTCOMES:
Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) | Baseline, 12 weeks after start of treatment and three month after treatment has ended.
  Diagnostic interview
Clinical Global Impression - Severity (CGI-S) | Baseline, 12 weeks after start of treatment and three month after treatment has ended.
  Clinician rated severity of symptoms
Clinical Global Impression - Improvement (CGI-I) | At 12 weeks after start of treatment and three month after treatment has ended.
  Clinician rated improvement after treatment
Children's Global Assessment Scale (CGAS) | Baseline, 12 weeks after start of treatment and three month after treatment has ended.
  Clinician rated global functioning
Brief Intolerance of Uncertainty Scale (Brief IUS) | Baseline, weekly during treatment, 12 weeks after treatment starts, and three months after treatment has ended
  Self rated tolerance to treatment
Brief Cognitive Avoidance Questionnaire (Brief CAQ) | Baseline, weekly during treatment, 12 weeks after treatment starts, and three months after treatment has ended
  Self rated cognitive avoidance
Brief Why Worry-II (Brief WW2) | Baseline, weekly during treatment, 12 weeks after treatment starts, and three months after treatment has ended
  Self rated positive assumptions of worry
Negative Problem Orientation Questionnaire (NPOQ) | Baseline, weekly during treatment, 12 weeks after treatment starts, and three months after treatment has ended
  Self rated negative problem orientation
Revised Children´s Anxiety and Depression Scale (RCADS-C) | Baseline, 12 weeks after start of treatment and three month after treatment has ended.
  Child and parent version.
Education, Work and Social Adjustment Scale (EWSAS) | Baseline, 12 weeks after start of treatment and three month after treatment has ended.
  Child and parent version.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No